CLINICAL TRIAL: NCT06432725
Title: Enhancing HIV Prevention and Treatment Referral and Engagement Among Latino Men Who Have Sex With Men (MSM): A Pilot Hybrid Effectiveness-Implementation Trial of the JUNTOS Referral Network
Brief Title: Joining Under-connected Networks to Optimize "Salud" (Health) ("JUNTOS")
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Audrey Harkness, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20230443; R34MH134670 (NIH)
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JUNTOS (Experimental): Participants in this group will get access to the JUNTOS Referral Network website/app through the 6-month follow up (HIV test counselors) and 3-month follow up (Latino MSM).
  Interventions: Behavioral: JUNTOS
- Referral Sheet - HIV test counselors (Active Comparator): Participants in this group will get access to the referral sheet through the 6-month follow up (HIV test counselors) and 3-month follow up (Latino MSM).
  Interventions: Behavioral: Referral Sheet

INTERVENTIONS:
Behavioral: JUNTOS — HIV test counselor and Latino MSM participants will be given access to the JUNTOS website/app, which shows information about local HIV and ancillary services. HIV test counselor participants will also be given access to a training video explaining how to use the JUNTOS website/app. HIV test counselors are encouraged to use the website/app for approximately 10 minutes at least once a week when meeting with Latino MSM testing clients. Latino MSM are encouraged to use the website/app to locate HIV and ancillary services as needed.
  Arms: JUNTOS
Behavioral: Referral Sheet — HIV test counselor and Latino MSM participants will be given access to referral sheet, which is a list of local HIV and ancillary services. HIV test counselors are encouraged to use the referral sheet for approximately 10 minutes at least once a week when meeting with Latino MSM testing clients. Latino MSM are encouraged to use the referral sheet to locate HIV and ancillary services as needed.
  Arms: Referral Sheet - HIV test counselors

SUMMARY:
The objective of this study is to evaluate the JUNTOS Referral Network as an implementation strategy to enhance the reach of HIV-prevention and treatment services to Latino gay, bisexual, and other men who have sex with men (MSM).

ELIGIBILITY:
Inclusion Criteria:

HIV Test counselors:

* 18 years of age or older
* Certified as an HIV test counselor in Miami-Dade County or Broward County (at the time of enrollment)
* Working or volunteering as an HIV test counselor in Miami-Dade County or Broward County and report testing 2 or more Latino MSM client per month (at the time of enrollment)
* Plans to continue working or volunteering as an HIV test counselor in Miami-Dade County or Broward County for the next 6 months
* Reports suboptimal fidelity to pre-exposure prophylaxis (PrEP) referral guidelines (<90% fidelity) and/or self-reports an unmet need for HIV prevention/treatment referral resources
* Willing and able to recruit up to 5 Latino MSM testing clients into the study

Latino MSM:

* 18 years of age or older
* Identifies as Latino/a/x or Hispanic
* Identifies as a sexual minority man or reports being a man who has sex with men
* Speaks English and/or Spanish
* Received an HIV test from an HIV test counselor participating in the study or completed an HIV test with a counselor in the last 3 months
* Lives in Miami-Dade County, Broward County, or Palm Beach County and anticipates living there for the next three months

Exclusion Criteria:

HIV test counselors:

* Unable to consent
* Study personnel unable to verify HIV test counselor role in Miami-Dade County or Broward County (e.g., confirmation of where they work/volunteer as HIV test counselor, location they state they provide services doesn't exist or does not provide HIV testing services)
* Works as an HIV test counselor in an incarceration/prison setting (i.e., clients are prisoners)

Latino MSM:

* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Use of Biomedical HIV Prevention/Treatment | 3-months
  The number of Latino MSM participants who indicated using a biomedical HIV prevention/treatment.
Percentage of Latino MSM Referral for Biomedical HIV Prevention/Treatment | 3-months
  The Referral Fidelity Questionnaire, developed for this study, has scores that range from 0% to 100%. Higher scores indicate more Latino MSM clients were referred to biomedical HIV Prevention/Treatment.

SECONDARY OUTCOMES:
Percentage of Latino MSM Referral for Biomedical HIV Prevention/Treatment | 6-months
  The Referral Fidelity Questionnaire, developed for this study, has scores that range from 0% to 100%. Higher scores indicate more Latino MSM clients referred to biomedical HIV Prevention/Treatment.
HIV acquisition, measures by self-report | 3-months
  This will be measured by a self-report question of Latino MSM's HIV status.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Harkness, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No